CLINICAL TRIAL: NCT04830904
Title: Efficacy of Lycra Garments in Ataxic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 760
Record Dates: First submitted 2021-03-11; First posted 2021-04-05 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ataxia, Cerebellar
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of lycra garments (Experimental): the subjects are assessed with and without wearing the device
  Interventions: Device: personalized Lycra garments

INTERVENTIONS:
Device: personalized Lycra garments — the subjects wear lycra garments during the assessment time and for some days after the assessment

SUMMARY:
The aim of this study iss to analyze the effect of Lycra garments in the axial stabilization in subjects affected by ataxia, both in acquired cerebellar injuries and malformative etiology.

Improvement are expected for what concerns:

* greater stability during stance
* smoother walking pattern
* reduction of risk of fall.

The two groups (acquired and malformative) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* subjects recruited must show a framework of ataxia consequent to acquired brain injury or malformative etiology.
* subjects must be able to walk autonomously without any device

Exclusion Criteria:

* presence of spasticity or muscular contractures
* subjects who already used lycra garments

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement of the center of mass over GRAIL/no device | immediately before wearing the lycra garment
  Balance in static conditions and Walking assessment over GRAIL. GRAIL will be used to track the movement of the Center Of Mass of the patient during 4 repetitions lasting 1 minute
Movement of the center of mass over GRAIL/ with lycra garments | immediately after wearing the lycra garment
  Balance in static conditions and Walking assessment over GRAIL. GRAIL will be used to track the movement of the Center Of Mass of the patient during 4 repetition lasting 1 minute
Berg Balance Scale/no device | immediately before wearing the lycra garment
  Berg Balance Scale is a scale to assess the risk of fall and balance failure. It ranges from 0 (worse outcome) to 56 (best outcome)
Berg Balance Scale/ with lycra garments | immediately after wearing the lycra garment
  Berg Balance Scale is a scale to assess the risk of fall and balance failure. It ranges from 0 (worse outcome) to 56 (best outcome)
6 Minute Walking Test/no device | immediately before wearing the lycra garment
  a test to assess the walking resistance
6 Minute Walking Test/ with lycra garments | immediately after wearing the lycra garment
  a test to assess the walking resistance
Goal Attainment Scaling/no device | immediately before wearing the device
  Goal Attainment Scaling is a subjective scale that can be defined between clinicians and subjects (or their parents) to identify changes in specific activities. It should be articulated up to 3 goals, and each of them should be scored with values ranging from -2 (worse score) to +2 (better)
Goal Attainment Scaling/ with lycra garments | immediately after wearing the lycra garment
  Goal Attainment Scaling is a subjective scale that can be defined between clinicians and subjects (or their parents) to identify changes in specific activities. It should be articulated up to 3 goals, and each of them should be scored with values ranging from -2 (worse score) to +2 (better)

SECONDARY OUTCOMES:
Likert tolerability questionaire | 14 days after wearing the lycra garment
  a likert tool designed to evaluate the tolerability of the lycra garments

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No